CLINICAL TRIAL: NCT02428374
Title: Role of Innate and Adaptive Immunity After Acute Myocardial Infarction BATTLE-AMI Study (B And T Types of Lymphocytes Evaluation in Acute Myocardial Infarction)
Brief Title: Role of Immune Responses After Acute Myocardial Infarction
Acronym: BATTLE-AMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Francisco Antonio Helfenstein Fonseca, Affiliate Professor of Medicine, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPM/UNIFESP; FAPESP (Other Grant/Funding Number: Research Foundation of the State of Sao Paulo)
Record Dates: First submitted 2015-03-10; First posted 2015-04-28 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Myocardial Fibrosis
Keywords: MRI; Ventricular function, left
MeSH Terms: interventions — Rosuvastatin Calcium; Clopidogrel; Ticagrelor; Simvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- rosuvastatin plus clopidogrel (Active Comparator): rosuvastatin 40 mg and clopidogrel 75 mg
  Interventions: Drug: Rosuvastatin plus ticagrelor; Drug: Simvastatin plus clopidogrel; Drug: Simvastatin plus ticagrelor
- Rosuvastatin plus ticagrelor (Active Comparator): Rosuvastatin 40 mg plus ticagrelor 90 mg bid
  Interventions: Drug: Rosuvastatin plus clopidogrel; Drug: Simvastatin plus clopidogrel; Drug: Simvastatin plus ticagrelor
- simvastatin plus clopidogrel (Active Comparator): Simvastatin 40 mg plus clopidogrel 75 mg
  Interventions: Drug: Rosuvastatin plus clopidogrel; Drug: Rosuvastatin plus ticagrelor; Drug: Simvastatin plus ticagrelor
- Simvastatin plus ticagrelor (Active Comparator): Simvastatin 40 mg plus ticagrelor 90 mg bid
  Interventions: Drug: Rosuvastatin plus clopidogrel; Drug: Rosuvastatin plus ticagrelor; Drug: Simvastatin plus clopidogrel

INTERVENTIONS:
Drug: Rosuvastatin plus clopidogrel — Crestor 40 mg daily plus Plavix 600 mg (initial dosis) and 75 mg daily up to 6-mo
  Other Names: Crestor & Plavix
  Arms: Rosuvastatin plus ticagrelor; Simvastatin plus ticagrelor; simvastatin plus clopidogrel
Drug: Rosuvastatin plus ticagrelor — Crestor 40 mg plus Brilinta 180 mg (initial dosis) and 90 mg bid up to 6-mo
  Other Names: Crestor & Brilinta
  Arms: Simvastatin plus ticagrelor; rosuvastatin plus clopidogrel; simvastatin plus clopidogrel
Drug: Simvastatin plus clopidogrel — Zocor 40 mg plus Plavix 600 mg (initial dosis) and 75 mg daily up to 6-mo
  Other Names: Zocor plus Plavix
  Arms: Rosuvastatin plus ticagrelor; Simvastatin plus ticagrelor; rosuvastatin plus clopidogrel
Drug: Simvastatin plus ticagrelor — Zocor 40 mg plus Brilinta 180 mg (initial dosis) and 90 mg bid up to 6-mo
  Other Names: Zocor & Brilinta
  Arms: Rosuvastatin plus ticagrelor; rosuvastatin plus clopidogrel; simvastatin plus clopidogrel

SUMMARY:
The fascinating role of lymphocyte subtypes in the development of coronary artery disease may be a new strategic target for understanding and therapy of acute myocardial infarction. The determinants of cell viability are unknown, postulating that they arise from factors not only related to microcirculation or energy expenditure, but also to inflammatory and immune responses. Furthermore, the intense mobilization of progenitor cells secondary to myocardial infarction triggers large lymphocyte proliferation that colonizes plaques in development, contributing to recurrent ischemic outcomes. This project aims to evaluate the immune and metabolic mechanisms involved in the recovery of the ischemic myocardium and coronary disease progression.

DETAILED DESCRIPTION:
Specifically, the investigators will study the innate and adaptive immunity, with emphasis on lymphocytes subtypes involved in the early and late surrogate outcomes of patients with acute myocardial infarction, their characterization (B1, B2 and T lymphocytes) in cell culture and by flow-cytometry, and immune responses (IgM and IgG for oxLDL and specific epitopes of apoB). In addition, the project will evaluate new biomarkers identified by studies of metabolomics, as well as the corresponding signaling pathways. Therapeutic pharmacological strategies and changes on intestinal microbiota will be evaluated since the acute phase of myocardial infarction up to 6 months.

In the study, the investigators will compared four arms of combined therapy: clopidogrel with rosuvastatin; or clopidogrel with simvastatin; or ticagrelor with rosuvastatin; or ticagrelor with simvastatin. The investigator's hypothesis is that the improvement of microcirculation with rosuvastatin and ticagrelor (synergic pleiotropic effects) may decrease the infarcted mass area, resulting in better left ventricular ejection fraction when compared to the other combined therapies.

The monitoring and genotype of microbiota will be examined together the metabolomics and cardiac MRIs obtained at the acute phase of MI and after 1-mo and 6-mo FU.

ELIGIBILITY:
Inclusion Criteria:

1. Stable patients with ST elevation myocardial infarction (STEMI) treated with thrombolytics in the first 6h or the initial of symptoms of MI.

Exclusion Criteria:

1. Contraindication or known intolerance to the study drug protocol
2. Those with comorbidities such as neoplasm, renal insufficiency (stage 4 or higher)

Patients should be randomized in the first 24 hours of AMI and treated by one of the four combined therapies at least 2h prior to coronary angiogram followed by percutaneous intervention when necessary.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-04 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of the left ventricular function (MRI) between the four combined treatments, after STEMI | 1-mo
  The effects of treatments on the left ventricular function will be measured by MRI

SECONDARY OUTCOMES:
To compare the effects of the four combined therapies on the left ventricular function after STEMI | 3-d
  Variables will be examined by MRI
To compare the effects of the four combined therapies on the left ventricular function after STEMI | 6-mo
  Variables will be examined by MRI
To compare the effects of the four combined therapies on the infarcted mass area after STEMI | 1-mo
  Variables will be examined by MRI
To compare the effects of the four combined therapies on the infarcted mass area after STEMI | 6-mo
  Variables will be examined by MRI
To compare the effects of the four combined therapies on the percentage of subjects with left ventricular ejection fraction < 40% after STEMI | 1-mo
  Variables will be examined by MRI
To compare the effects of the four combined therapies on the percentage of subjects with left ventricular ejection fraction < 40% after STEMI | 6-mo
  Variables will be examined by MRI
To quantify the percentage and absolute number of B1, B2, TCD4, and TCD8 subtypes of lymphocytes and their correlation with left ventricular ejection fraction after STEMI | 1-d
  Lymphocyte subtypes quantified by flow-cytometry and left ventricular ejection fraction by MRI
To quantify the percentage and absolute number of B1, B2, TCD4, and TCD8 subtypes of lymphocytes and their correlation with left ventricular ejection fraction after STEMI | 1-mo
  Lymphocyte subtypes quantified by flow-cytometry and left ventricular ejection fraction by MRI
To quantify the percentage and absolute number of B1, B2, TCD4, and TCD8 subtypes of lymphocytes and their correlation with left ventricular ejection fraction after STEMI | 6-mo
  Lymphocyte subtypes quantified by flow-cytometry and left ventricular ejection fraction by MRI
To quantify the percentage and absolute number of B1, B2, TCD4, and TCD8 subtypes of lymphocytes and their correlation with infarcted mass area after STEMI | 1-d
  Lymphocyte subtypes quantified by flow-cytometry and infarcted mass area by MRI
To quantify the percentage and absolute number of B1, B2, TCD4, and TCD8 subtypes of lymphocytes and their correlation with infarcted mass area after STEMI | 1-mo
  Lymphocyte subtypes quantified by flow-cytometry and infarcted mass area by MRI
To quantify the percentage and absolute number of B1, B2, TCD4, and TCD8 subtypes of lymphocytes and their correlation with infarcted mass area after STEMI | 6-mo
  Lymphocyte subtypes quantified by flow-cytometry and infarcted mass area by MRI
To quantify the percentage and absolute number of B1, B2, TCD4, and TCD8 subtypes of lymphocytes and their correlation with left ventricular ejection fraction <40% after STEMI | 1-d
  Lymphocyte subtypes quantified by flow-cytometry and left ventricular ejection fraction by MRI
To quantify the percentage and absolute number of B1, B2, TCD4, and TCD8 subtypes of lymphocytes and their correlation with left ventricular ejection fraction <40% after STEMI | 1-mo
  Lymphocyte subtypes quantified by flow-cytometry and left ventricular ejection fraction by MRI
To quantify the percentage and absolute number of B1, B2, TCD4, and TCD8 subtypes of lymphocytes and their correlation with left ventricular ejection fraction <40% after STEMI | 6-mo
  Lymphocyte subtypes quantified by flow-cytometry and left ventricular ejection fraction by MRI

OTHER OUTCOMES:
Relationship between gut microbiota and diabetes status after STEMI | 1-3d
  Intestinal microbiota will be genotyped and diabetes status (non-diabetic, pre-diabetic or diabetic) according to HbA1c levels.
Relationship between gut microbiota and diabetes status after STEMI | 1-mo
  Intestinal microbiota will be genotyped and diabetes status (non-diabetic, pre-diabetic or diabetic) according to HbA1c levels.
Relationship between gut microbiota and diabetes status | 6-mo
  Intestinal microbiota will be genotyped and diabetes status (non-diabetic, pre-diabetic or diabetic) according to HbA1c levels.
Relationship between gut microbiota and metabolomics | 1-3d
  Intestinal microbiota will be genotyped and metabolomics by LC/MS-MS
Relationship between gut microbiota and metabolomics | 1-mo
  Intestinal microbiota will be genotyped and metabolomics by LC/MS-MS
Relationship between gut microbiota and metabolomics | 6-mo
  Intestinal microbiota will be genotyped and metabolomics by LC/MS-MS
Comparison between the four arm of combined therapies on microparticles and endothelial progenitor cells | 1-d
  Endothelial, platelet, and monocyte-derived microparticles as well as endothelial progenitor cells will be quantified by flow-cytometry
Comparison between the four arm of combined therapies on microparticles and endothelial progenitor cells | 1-mo
  Endothelial, platelet, and monocyte-derived microparticles as well as endothelial progenitor cells will be quantified by flow-cytometry
Comparison between the four arm of combined therapies on microparticles and endothelial progenitor cells | 6-mo
  Endothelial, platelet, and monocyte-derived microparticles as well as endothelial progenitor cells will be quantified by flow-cytometry
Correlation between the severity of coronary disease with antibodies against oxidized LDL and peptide D of apolipoprotein B of LDL | 1-d
  Antibodies IgG and IgM against oxidized LDL as well as against peptide D of LDL will be quantified by ELISA. Coronary disease severity will be quantified by the Gensini Score
Comparison between the four arms of combined therapies on TIMI flow grade and blush grade | 1-d
  TIMI flow grade and blush grade will be determined based on coronary angiogram obtained at baseline by two independent and blinded certified invasive cardiologists
Relationship between no-reflow images obtained at MRI with metabolomics | 1-d
  Metabolomics will be determined by LC/MS-MS and images by MRI
Relationship between no-reflow images obtained at MRI with metabolomics | 1-mo
  Metabolomics will be determined by LC/MS-MS and images by MRI
Relationship between no-reflow images obtained at MRI with metabolomics | 6-mo
  Metabolomics will be determined by LC/MS-MS and images by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Francisco A Fonseca, MD, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Hospital Sao Paulo - UNIFESP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Fonseca FA, Izar MC, Fuster V, Gallo R, Padurean A, Fallon JT, Schachter EN, Chesebro JH, Badimon JJ. Chronic endothelial dysfunction after oversized coronary balloon angioplasty in pigs: a 12-week follow-up of coronary vasoreactivity in vivo and in vitro. Atherosclerosis. 2001 Jan;154(1):61-9. doi: 10.1016/s0021-9150(00)00458-5. PMID 11137083
- [Background] Silva EP, Fonseca FA, Ihara SS, Izar MC, Lopes IL, Pinto LE, Badimon JJ, Tuffik S, Paiva TB, Kasinski N, de Paola AV, Carvalho AC. Early benefits of pravastatin to experimentally induced atherosclerosis. J Cardiovasc Pharmacol. 2002 Mar;39(3):389-95. doi: 10.1097/00005344-200203000-00010. PMID 11862118
- [Background] Fonseca FA, Paiva TB, Silva EG, Ihara SS, Kasinski N, Martinez TL, Filho EE. Dietary magnesium improves endothelial dependent relaxation of balloon injured arteries in rats. Atherosclerosis. 1998 Aug;139(2):237-42. doi: 10.1016/s0021-9150(98)00069-0. PMID 9712329
- [Background] Fonseca FA, Ihara SS, Izar MC, Silva EP, Kasinski N, Lopes IE, Pinto LE, Paiva TB, Tufik S, de Paola AA, Carvalho AC. Hydrochlorothiazide abolishes the anti-atherosclerotic effect of quinapril. Clin Exp Pharmacol Physiol. 2003 Oct;30(10):779-85. doi: 10.1046/j.1440-1681.2003.03911.x. PMID 14516418
- [Background] Ferreira WP, Bertolami MC, Santos SN, Barros MR, de Matos Barretto RB, Pontes SC Jr, Fonseca FH, Carvalho AC. One-month therapy with simvastatin restores endothelial function in hypercholesterolemic children and adolescents. Pediatr Cardiol. 2007 Jan-Feb;28(1):8-13. doi: 10.1007/s00246-005-1304-x. Epub 2007 Jan 25. PMID 17318708
- [Background] Monteiro CM, Pinheiro LF, Izar MC, Barros SW, Vasco MB, Fischer SM, Povoa RM, Brandao SA, Santos AO, Oliveira L, Carvalho AC, Fonseca FA. Highly sensitive C-reactive protein and male gender are independently related to the severity of coronary disease in patients with metabolic syndrome and an acute coronary event. Braz J Med Biol Res. 2010 Mar;43(3):297-302. doi: 10.1590/s0100-879x2010005000008. Epub 2010 Mar 5. PMID 20209376
- [Background] da Silva EF, Fonseca FA, Franca CN, Ferreira PR, Izar MC, Salomao R, Camargo LM, Tenore SB, Lewi DS. Imbalance between endothelial progenitors cells and microparticles in HIV-infected patients naive for antiretroviral therapy. AIDS. 2011 Aug 24;25(13):1595-601. doi: 10.1097/QAD.0b013e32834980f4. PMID 21673561
- [Background] Franca CN, Pinheiro LF, Izar MC, Brunialti MK, Salomao R, Bianco HT, Kasmas SH, Barbosa SP, de Nucci G, Fonseca FA. Endothelial progenitor cell mobilization and platelet microparticle release are influenced by clopidogrel plasma levels in stable coronary artery disease. Circ J. 2012;76(3):729-36. doi: 10.1253/circj.cj-11-1145. Epub 2011 Dec 28. PMID 22214900
- [Background] Pomaro DR, Ihara SS, Pinto LE, Ueda I, Casarini DE, Ebihara F, Santos AO, Izar MC, Fonseca FA. High glucose levels abolish antiatherosclerotic benefits of ACE inhibition in alloxan-induced diabetes in rabbits. J Cardiovasc Pharmacol. 2005 Apr;45(4):295-300. doi: 10.1097/01.fjc.0000155384.64350.45. PMID 15772516
- [Background] Relvas WG, Izar MC, Segreto HR, Giordani AJ, Ihara SS, Mariano M, Lopes JD, Popi AF, Helfenstein T, Pomaro D, Povoa RM, Carvalho AC, Fonseca FA. Resident peritoneal inflammatory cells are pivotal in the development of experimental atherosclerosis. J Atheroscler Thromb. 2010 Apr 30;17(4):378-85. doi: 10.5551/jat.3418. Epub 2010 Mar 9. PMID 20215709
- [Background] Helfenstein T, Fonseca FA, Ihara SS, Bottos JM, Moreira FT, Pott H Jr, Farah ME, Martins MC, Izar MC. Impaired glucose tolerance plus hyperlipidaemia induced by diet promotes retina microaneurysms in New Zealand rabbits. Int J Exp Pathol. 2011 Feb;92(1):40-9. doi: 10.1111/j.1365-2613.2010.00753.x. PMID 21272105
- [Background] Feio CA, Izar MC, Ihara SS, Kasmas SH, Martins CM, Feio MN, Maues LA, Borges NC, Moreno RA, Povoa RM, Fonseca FA. Euterpe oleracea (acai) modifies sterol metabolism and attenuates experimentally-induced atherosclerosis. J Atheroscler Thromb. 2012;19(3):237-45. doi: 10.5551/jat.11205. Epub 2011 Dec 3. PMID 22139433
- [Background] Albert MA, Glynn RJ, Fonseca FA, Lorenzatti AJ, Ferdinand KC, MacFadyen JG, Ridker PM. Race, ethnicity, and the efficacy of rosuvastatin in primary prevention: the Justification for the Use of Statins in Prevention: an Intervention Trial Evaluating Rosuvastatin (JUPITER) trial. Am Heart J. 2011 Jul;162(1):106-14.e2. doi: 10.1016/j.ahj.2011.03.032. Epub 2011 Jun 12. PMID 21742096
- [Background] de Lima Sanches P, de Mello MT, Elias N, Fonseca FA, de Piano A, Carnier J, Oyama LM, Tock L, Tufik S, Damaso AR. Improvement in HOMA-IR is an independent predictor of reduced carotid intima-media thickness in obese adolescents participating in an interdisciplinary weight-loss program. Hypertens Res. 2011 Feb;34(2):232-8. doi: 10.1038/hr.2010.225. Epub 2010 Dec 2. PMID 21124323
- [Background] Fonseca FA, Franca CN, Povoa RM, Izar MC. [Statins and stroke: potential mechanisms for neurovascular protection]. Rev Neurol. 2010 Nov 1;51(9):551-60. Spanish. PMID 20979035
- [Background] Ridker PM, MacFadyen JG, Fonseca FA, Genest J, Gotto AM, Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, Nordestgaard BG, Shepherd J, Willerson JT, Glynn RJ; JUPITER Study Group. Number needed to treat with rosuvastatin to prevent first cardiovascular events and death among men and women with low low-density lipoprotein cholesterol and elevated high-sensitivity C-reactive protein: justification for the use of statins in prevention: an intervention trial evaluating rosuvastatin (JUPITER). Circ Cardiovasc Qual Outcomes. 2009 Nov;2(6):616-23. doi: 10.1161/CIRCOUTCOMES.109.848473. Epub 2009 Sep 22. PMID 20031900
- [Background] Brandao SA, Izar MC, Fischer SM, Santos AO, Monteiro CM, Povoa RM, Helfenstein T, Carvalho AC, Monteiro AM, Ramos E, Gidlund M, Figueiredo Neto AM, Fonseca FA. Early increase in autoantibodies against human oxidized low-density lipoprotein in hypertensive patients after blood pressure control. Am J Hypertens. 2010 Feb;23(2):208-14. doi: 10.1038/ajh.2009.214. Epub 2009 Nov 12. PMID 19910928
- [Background] Fonseca FA, Izar MC. Primary prevention of vascular events in patients with high levels of C-reactive protein: the JUPITER study. Expert Rev Cardiovasc Ther. 2009 Sep;7(9):1041-56. doi: 10.1586/erc.09.93. PMID 19764857
- [Background] Santos AO, Fonseca FA, Fischer SM, Monteiro CM, Brandao SA, Povoa RM, Bombig MT, Carvalho AC, Monteiro AM, Ramos E, Gidlund M, Figueiredo Neto AM, Izar MC. High circulating autoantibodies against human oxidized low-density lipoprotein are related to stable and lower titers to unstable clinical situation. Clin Chim Acta. 2009 Aug;406(1-2):113-8. doi: 10.1016/j.cca.2009.06.005. Epub 2009 Jun 10. PMID 19523463
- [Background] Glynn RJ, Danielson E, Fonseca FA, Genest J, Gotto AM Jr, Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, MacFadyen JG, Nordestgaard BG, Shepherd J, Willerson JT, Ridker PM. A randomized trial of rosuvastatin in the prevention of venous thromboembolism. N Engl J Med. 2009 Apr 30;360(18):1851-61. doi: 10.1056/NEJMoa0900241. Epub 2009 Mar 29. PMID 19329822
- [Background] Ridker PM, Danielson E, Fonseca FA, Genest J, Gotto AM Jr, Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, Macfadyen JG, Nordestgaard BG, Shepherd J, Willerson JT, Glynn RJ; JUPITER Trial Study Group. Reduction in C-reactive protein and LDL cholesterol and cardiovascular event rates after initiation of rosuvastatin: a prospective study of the JUPITER trial. Lancet. 2009 Apr 4;373(9670):1175-82. doi: 10.1016/S0140-6736(09)60447-5. Epub 2009 Mar 28. PMID 19329177
- [Background] Ridker PM, Danielson E, Fonseca FA, Genest J, Gotto AM Jr, Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, MacFadyen JG, Nordestgaard BG, Shepherd J, Willerson JT, Glynn RJ; JUPITER Study Group. Rosuvastatin to prevent vascular events in men and women with elevated C-reactive protein. N Engl J Med. 2008 Nov 20;359(21):2195-207. doi: 10.1056/NEJMoa0807646. Epub 2008 Nov 9. PMID 18997196
- [Background] Ridker PM, Fonseca FA, Genest J, Gotto AM, Kastelein JJ, Khurmi NS, Koenig W, Libby P, Lorenzatti AJ, Nordestgaard BG, Shepherd J, Willerson JT, Glynn RJ; JUPITER Trial Study Group. Baseline characteristics of participants in the JUPITER trial, a randomized placebo-controlled primary prevention trial of statin therapy among individuals with low low-density lipoprotein cholesterol and elevated high-sensitivity C-reactive protein. Am J Cardiol. 2007 Dec 1;100(11):1659-64. doi: 10.1016/j.amjcard.2007.09.072. Epub 2007 Oct 24. PMID 18036365
- [Background] Ramos SC, Fonseca FA, Kasmas SH, Moreira FT, Helfenstein T, Borges NC, Moreno RA, Rezende VM, Silva FC, Izar MC. The role of soluble fiber intake in patients under highly effective lipid-lowering therapy. Nutr J. 2011 Aug 2;10:80. doi: 10.1186/1475-2891-10-80. PMID 21810257
- [Background] Izar MC, Tegani DM, Kasmas SH, Fonseca FA. Phytosterols and phytosterolemia: gene-diet interactions. Genes Nutr. 2011 Feb;6(1):17-26. doi: 10.1007/s12263-010-0182-x. Epub 2010 Aug 28. PMID 21437027
- [Background] Fonseca HA, Izar MC, Bianco HT, Fonseca FA. Ezetimibe, oxidized low density lipoprotein, Lp (a), and dyslipidemia. J Atheroscler Thromb. 2010 Aug 31;17(8):888. doi: 10.5551/jat.5918. Epub 2010 Aug 10. No abstract available. PMID 20702973
- [Background] Kasmas SH, Izar MC, Franca CN, Ramos SC, Moreira FT, Helfenstein T, Moreno RA, Borges NC, Figueiredo-Neto AM, Fonseca FA. Differences in synthesis and absorption of cholesterol of two effective lipid-lowering therapies. Braz J Med Biol Res. 2012 Nov;45(11):1095-101. doi: 10.1590/s0100-879x2012007500118. Epub 2012 Jul 19. PMID 22801416
- [Background] da Fonseca HA, Fonseca FA, Monteiro AM, Farias NC Jr, Bianco HT, Brandao SA, Povoa RM, Gidlund M, Izar MC. Inflammatory environment and immune responses to oxidized LDL are linked to systolic and diastolic blood pressure levels in hypertensive subjects. Int J Cardiol. 2012 May 17;157(1):131-3. doi: 10.1016/j.ijcard.2012.03.041. Epub 2012 Mar 28. No abstract available. PMID 22459380
- [Background] Izar MC, Fonseca HA, Pinheiro LF, Monteiro CM, Povoa RM, Monteiro AM, Figueiredo-Neto AM, Gidlund MA, Fonseca FA. Adaptive immunity is related to coronary artery disease severity after acute coronary syndrome in subjects with metabolic syndrome. Diab Vasc Dis Res. 2013 Jan;10(1):32-9. doi: 10.1177/1479164112443374. Epub 2012 Apr 23. PMID 22529217
- [Background] Colossimo AP, Costa Fde A, Riera AR, Bombig MT, Lima VC, Fonseca FA, Izar MC, L Filho B, Souza D, Povoa RM. Electrocardiogram sensitivity in left ventricular hypertrophy according to gender and cardiac mass. Arq Bras Cardiol. 2011 Sep;97(3):225-31. doi: 10.1590/s0066-782x2011005000085. Epub 2011 Aug 12. English, Portuguese. PMID 21845342
- [Background] Costa Fde A, Bombig MT, de Lima VC, de Souza D, Luna Filho B, Fonseca FH, Izar MC, da Costa W, Riera AR, Povoa R. Geometric patterns of left ventricular hypertrophy and electrocardiography. Int J Cardiol. 2011 Sep 15;151(3):374-5. doi: 10.1016/j.ijcard.2011.06.103. Epub 2011 Jul 18. No abstract available. PMID 21764471
- [Background] Marui FR, Bombig MT, Francisco YA, Thalenberg JM, Fonseca FA, Souza Dd, Costa Fde A, Izar MC, Carvalho AC, Povoa R. [Assessment of resistant hypertension with home blood pressure monitoring]. Arq Bras Cardiol. 2010 Oct;95(4):536-40. doi: 10.1590/s0066-782x2010005000120. Epub 2010 Sep 8. Multiple languages. PMID 20835685
- [Background] Santos MA, Costa Fde A, Travessa AF, Bombig MT, Fonseca FH, Luna Filho B, Mussi A, Souza Dd, Oliveira Ad, Povoa R. [Duchenne muscular dystrophy: electrocardiographic analysis of 131 patients]. Arq Bras Cardiol. 2010 May;94(5):620-4. doi: 10.1590/s0066-782x2010005000024. Epub 2010 Apr 2. Portuguese. PMID 20379617
- [Background] Schwartz GG, Olsson AG, Ballantyne CM, Barter PJ, Holme IM, Kallend D, Leiter LA, Leitersdorf E, McMurray JJ, Shah PK, Tardif JC, Chaitman BR, Duttlinger-Maddux R, Mathieson J; dal-OUTCOMES Committees and Investigators. Rationale and design of the dal-OUTCOMES trial: efficacy and safety of dalcetrapib in patients with recent acute coronary syndrome. Am Heart J. 2009 Dec;158(6):896-901.e3. doi: 10.1016/j.ahj.2009.09.017. PMID 19958854
- [Background] Brollo L, Bombig MT, Mazzaro Cdo L, Francisco YA, Fonseca FA, Carvalho AC, Harima H, Hirai A, Povoa R. Relationship between electrocardiogram with diabetes mellitus and metabolic syndrome in Japanese-Brazilians. Arq Bras Cardiol. 2009 May;92(5):351-5, 381-6. doi: 10.1590/s0066-782x2009000500008. English, Multiple languages. PMID 19629290
- [Background] Monteiro CM, Oliveira L, Izar MC, Helfenstein T, Santos AO, Fischer SM, Barros SW, Pinheiro LF, Carvalho AC, Fonseca FA. Early glucometabolic profile in patients with acute coronary syndromes and metabolic syndrome. Arq Bras Cardiol. 2009 Feb;92(2):89-99. doi: 10.1590/s0066-782x2009000200004. English, Portuguese, Spanish. PMID 19360240
- [Background] da Costa W, Riera AR, Costa Fde A, Bombig MT, de Paola AA, Carvalho AC, Fonseca FH, Luna Filho B, Povoa R. Correlation of electrocardiographic left ventricular hypertrophy criteria with left ventricular mass by echocardiogram in obese hypertensive patients. J Electrocardiol. 2008 Nov-Dec;41(6):724-9. doi: 10.1016/j.jelectrocard.2008.05.010. PMID 18954613
- [Background] Izar MC, Helfenstein T, Ihara SS, Relvas WG, Santos AO, Fischer SC, Pinto LE, Lopes IE, Pomaro DR, Fonseca MI, Bodanese LC, Moriguchi EH, Saraiva JF, Introcaso L, Souza AD, Scartezini M, Torres KP, Zagury L, Jardim PC, Costa EA, Tacito LH, Forti A, Magalhaes ME, Chacra AR, Bertolami MC, Loures-Vale AA, Barros MA, Xavier HT, Lyra R, Argamanijan D, Guimaraes A, Novazzi JP, Kasinski N, Afiune A, Martinez TL, Santos RD, Nicolau JC, Cesar LA, Povoa RM, Carvalho AC, Han SW, Fonseca FA; GOLD Investigators. Association of lipoprotein lipase D9N polymorphism with myocardial infarction in type 2 diabetes: the genetics, outcomes, and lipids in type 2 diabetes (GOLD) study. Atherosclerosis. 2009 May;204(1):165-70. doi: 10.1016/j.atherosclerosis.2008.08.006. Epub 2008 Aug 14. PMID 18823627
- [Background] Middleton A, Binbrek AS, Fonseca FA, Wilpshaar W, Watkins C, Strandberg TE. Achieving 2003 European lipid goals with rosuvastatin and comparator statins in 6743 patients in real-life clinical practice: DISCOVERY meta-analysis. Curr Med Res Opin. 2006 Jun;22(6):1181-91. doi: 10.1185/030079906X100177. PMID 16846551
- [Background] Helfenstein T, Fonseca FA, Relvas WG, Santos AO, Dabela ML, Matheus SC, D'Almeida V, Tufik S, Souza FG, Rodrigues PR, Taglieri R, Sousa EF, Izar MC. Prevalence of myocardial infarction is related to hyperhomocysteinemia but not influenced by C677T methylenetetrahydrofolate reductase and A2756G methionine synthase polymorphisms in diabetic and non-diabetic subjects. Clin Chim Acta. 2005 May;355(1-2):165-72. doi: 10.1016/j.cccn.2004.12.002. PMID 15820491
- [Background] Relvas WG, Izar MC, Helfenstein T, Fonseca MI, Colovati M, Oliveira A, Ihara SS, Han SW, Las Casas AA Jr, Fonseca FA. Relationship between gene polymorphisms and prevalence of myocardial infarction among diabetic and non-diabetic subjects. Atherosclerosis. 2005 Jan;178(1):101-5. doi: 10.1016/j.atherosclerosis.2004.05.025. PMID 15585206
- [Background] Pinheiro LF, Franca CN, Izar MC, Barbosa SP, Bianco HT, Kasmas SH, Mendes GD, Povoa RM, Fonseca FA. Pharmacokinetic interactions between clopidogrel and rosuvastatin: effects on vascular protection in subjects with coronary heart disease. Int J Cardiol. 2012 Jun 28;158(1):125-9. doi: 10.1016/j.ijcard.2012.04.051. Epub 2012 May 7. No abstract available. PMID 22569318
- [Background] Moore KJ, Tabas I. Macrophages in the pathogenesis of atherosclerosis. Cell. 2011 Apr 29;145(3):341-55. doi: 10.1016/j.cell.2011.04.005. PMID 21529710
- [Background] Weber C, Meiler S, Doring Y, Koch M, Drechsler M, Megens RT, Rowinska Z, Bidzhekov K, Fecher C, Ribechini E, van Zandvoort MA, Binder CJ, Jelinek I, Hristov M, Boon L, Jung S, Korn T, Lutz MB, Forster I, Zenke M, Hieronymus T, Junt T, Zernecke A. CCL17-expressing dendritic cells drive atherosclerosis by restraining regulatory T cell homeostasis in mice. J Clin Invest. 2011 Jul;121(7):2898-910. doi: 10.1172/JCI44925. PMID 21633167
- [Background] Vitale G, Mion F, Pucillo C. Regulatory B cells: evidence, developmental origin and population diversity. Mol Immunol. 2010 Nov-Dec;48(1-3):1-8. doi: 10.1016/j.molimm.2010.09.010. Epub 2010 Oct 14. PMID 20950861
- [Background] Miller YI, Choi SH, Wiesner P, Fang L, Harkewicz R, Hartvigsen K, Boullier A, Gonen A, Diehl CJ, Que X, Montano E, Shaw PX, Tsimikas S, Binder CJ, Witztum JL. Oxidation-specific epitopes are danger-associated molecular patterns recognized by pattern recognition receptors of innate immunity. Circ Res. 2011 Jan 21;108(2):235-48. doi: 10.1161/CIRCRESAHA.110.223875. PMID 21252151
- [Background] Galkina E, Kadl A, Sanders J, Varughese D, Sarembock IJ, Ley K. Lymphocyte recruitment into the aortic wall before and during development of atherosclerosis is partially L-selectin dependent. J Exp Med. 2006 May 15;203(5):1273-82. doi: 10.1084/jem.20052205. Epub 2006 May 8. PMID 16682495
- [Background] Ponnuswamy P, Van Vre EA, Mallat Z, Tedgui A. Humoral and cellular immune responses in atherosclerosis: spotlight on B- and T-cells. Vascul Pharmacol. 2012 May-Jun;56(5-6):193-203. doi: 10.1016/j.vph.2012.01.009. Epub 2012 Feb 8. PMID 22329947
- [Background] van Gils JM, Derby MC, Fernandes LR, Ramkhelawon B, Ray TD, Rayner KJ, Parathath S, Distel E, Feig JL, Alvarez-Leite JI, Rayner AJ, McDonald TO, O'Brien KD, Stuart LM, Fisher EA, Lacy-Hulbert A, Moore KJ. The neuroimmune guidance cue netrin-1 promotes atherosclerosis by inhibiting the emigration of macrophages from plaques. Nat Immunol. 2012 Jan 8;13(2):136-43. doi: 10.1038/ni.2205. PMID 22231519
- [Background] Campbell KA, Lipinski MJ, Doran AC, Skaflen MD, Fuster V, McNamara CA. Lymphocytes and the adventitial immune response in atherosclerosis. Circ Res. 2012 Mar 16;110(6):889-900. doi: 10.1161/CIRCRESAHA.111.263186. PMID 22427326
- [Background] Gerszten RE, Tager AM. The monocyte in atherosclerosis--should I stay or should I go now? N Engl J Med. 2012 May 3;366(18):1734-6. doi: 10.1056/NEJMcibr1200164. No abstract available. PMID 22551134
- [Background] Goodchild TT, Robinson KA, Pang W, Tondato F, Cui J, Arrington J, Godwin L, Ungs M, Carlesso N, Weich N, Poznansky MC, Chronos NA. Bone marrow-derived B cells preserve ventricular function after acute myocardial infarction. JACC Cardiovasc Interv. 2009 Oct;2(10):1005-16. doi: 10.1016/j.jcin.2009.08.010. PMID 19850263
- [Background] Dutta P, Courties G, Wei Y, Leuschner F, Gorbatov R, Robbins CS, Iwamoto Y, Thompson B, Carlson AL, Heidt T, Majmudar MD, Lasitschka F, Etzrodt M, Waterman P, Waring MT, Chicoine AT, van der Laan AM, Niessen HW, Piek JJ, Rubin BB, Butany J, Stone JR, Katus HA, Murphy SA, Morrow DA, Sabatine MS, Vinegoni C, Moskowitz MA, Pittet MJ, Libby P, Lin CP, Swirski FK, Weissleder R, Nahrendorf M. Myocardial infarction accelerates atherosclerosis. Nature. 2012 Jul 19;487(7407):325-9. doi: 10.1038/nature11260. PMID 22763456
- [Background] Moreira FT, Ramos SC, Monteiro AM, Helfenstein T, Gidlund M, Damasceno NR, Neto AM, Izar MC, Fonseca FA. Effects of two lipid lowering therapies on immune responses in hyperlipidemic subjects. Life Sci. 2014 Mar 11;98(2):83-7. doi: 10.1016/j.lfs.2014.01.001. Epub 2014 Jan 18. PMID 24447629
- [Background] Hilgendorf I, Theurl I, Gerhardt LM, Robbins CS, Weber GF, Gonen A, Iwamoto Y, Degousee N, Holderried TA, Winter C, Zirlik A, Lin HY, Sukhova GK, Butany J, Rubin BB, Witztum JL, Libby P, Nahrendorf M, Weissleder R, Swirski FK. Innate response activator B cells aggravate atherosclerosis by stimulating T helper-1 adaptive immunity. Circulation. 2014 Apr 22;129(16):1677-87. doi: 10.1161/CIRCULATIONAHA.113.006381. Epub 2014 Jan 31. PMID 24488984
- [Background] Kyaw T, Tay C, Krishnamurthi S, Kanellakis P, Agrotis A, Tipping P, Bobik A, Toh BH. B1a B lymphocytes are atheroprotective by secreting natural IgM that increases IgM deposits and reduces necrotic cores in atherosclerotic lesions. Circ Res. 2011 Sep 30;109(8):830-40. doi: 10.1161/CIRCRESAHA.111.248542. Epub 2011 Aug 25. PMID 21868694
- [Background] Schwartz GG, Olsson AG, Ezekowitz MD, Ganz P, Oliver MF, Waters D, Zeiher A, Chaitman BR, Leslie S, Stern T; Myocardial Ischemia Reduction with Aggressive Cholesterol Lowering (MIRACL) Study Investigators. Effects of atorvastatin on early recurrent ischemic events in acute coronary syndromes: the MIRACL study: a randomized controlled trial. JAMA. 2001 Apr 4;285(13):1711-8. doi: 10.1001/jama.285.13.1711. PMID 11277825
- [Background] Cannon CP, Braunwald E, McCabe CH, Rader DJ, Rouleau JL, Belder R, Joyal SV, Hill KA, Pfeffer MA, Skene AM; Pravastatin or Atorvastatin Evaluation and Infection Therapy-Thrombolysis in Myocardial Infarction 22 Investigators. Intensive versus moderate lipid lowering with statins after acute coronary syndromes. N Engl J Med. 2004 Apr 8;350(15):1495-504. doi: 10.1056/NEJMoa040583. Epub 2004 Mar 8. PMID 15007110
- [Background] Spencer FA, Fonarow GC, Frederick PD, Wright RS, Every N, Goldberg RJ, Gore JM, Dong W, Becker RC, French W; National Registry of Myocardial Infarction. Early withdrawal of statin therapy in patients with non-ST-segment elevation myocardial infarction: national registry of myocardial infarction. Arch Intern Med. 2004 Oct 25;164(19):2162-8. doi: 10.1001/archinte.164.19.2162. PMID 15505131
- [Background] Fonarow GC, Wright RS, Spencer FA, Fredrick PD, Dong W, Every N, French WJ; National Registry of Myocardial Infarction 4 Investigators. Effect of statin use within the first 24 hours of admission for acute myocardial infarction on early morbidity and mortality. Am J Cardiol. 2005 Sep 1;96(5):611-6. doi: 10.1016/j.amjcard.2005.04.029. PMID 16125480
- [Background] Wright RS, Bybee K, Miller WL, Laudon DA, Murphy JG, Jaffe AS. Reduced risks of death and CHF are associated with statin therapy administered acutely within the first 24 h of AMI. Int J Cardiol. 2006 Apr 14;108(3):314-9. doi: 10.1016/j.ijcard.2005.05.014. Epub 2005 Jun 22. PMID 15975672
- [Background] Di Sciascio G, Patti G, Pasceri V, Gaspardone A, Colonna G, Montinaro A. Efficacy of atorvastatin reload in patients on chronic statin therapy undergoing percutaneous coronary intervention: results of the ARMYDA-RECAPTURE (Atorvastatin for Reduction of Myocardial Damage During Angioplasty) Randomized Trial. J Am Coll Cardiol. 2009 Aug 4;54(6):558-65. doi: 10.1016/j.jacc.2009.05.028. Epub 2009 Jul 2. PMID 19643320
- [Background] Yun KH, Oh SK, Rhee SJ, Yoo NJ, Kim NH, Jeong JW. 12-month follow-up results of high dose rosuvastatin loading before percutaneous coronary intervention in patients with acute coronary syndrome. Int J Cardiol. 2011 Jan 7;146(1):68-72. doi: 10.1016/j.ijcard.2010.04.052. Epub 2010 May 14. PMID 20471117
- [Background] Gurbel PA, Bliden KP, Butler K, Tantry US, Gesheff T, Wei C, Teng R, Antonino MJ, Patil SB, Karunakaran A, Kereiakes DJ, Parris C, Purdy D, Wilson V, Ledley GS, Storey RF. Randomized double-blind assessment of the ONSET and OFFSET of the antiplatelet effects of ticagrelor versus clopidogrel in patients with stable coronary artery disease: the ONSET/OFFSET study. Circulation. 2009 Dec 22;120(25):2577-85. doi: 10.1161/CIRCULATIONAHA.109.912550. Epub 2009 Nov 18. PMID 19923168
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] Wiviott SD, Braunwald E, McCabe CH, Montalescot G, Ruzyllo W, Gottlieb S, Neumann FJ, Ardissino D, De Servi S, Murphy SA, Riesmeyer J, Weerakkody G, Gibson CM, Antman EM; TRITON-TIMI 38 Investigators. Prasugrel versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2007 Nov 15;357(20):2001-15. doi: 10.1056/NEJMoa0706482. Epub 2007 Nov 4. PMID 17982182
- [Background] Serebruany VL. Mortality benefit in PLATO cannot be explained by antiplatelet properties of ticagrelor. Cardiology. 2010;117(3):231-3. doi: 10.1159/000322789. Epub 2011 Jan 5. PMID 21212672
- [Background] Serebruany VL. The TRITON versus PLATO trials: differences beyond platelet inhibition. Thromb Haemost. 2010 Feb;103(2):259-61. doi: 10.1160/TH09-10-0695. Epub 2009 Dec 18. PMID 20024505
- [Background] Serebruany VL, Atar D. The PLATO trial: do you believe in magic? Eur Heart J. 2010 Apr;31(7):764-7. doi: 10.1093/eurheartj/ehp545. Epub 2009 Dec 10. PMID 20007979
- [Background] Grzesk G, Kozinski M, Navarese EP, Krzyzanowski M, Grzesk E, Kubica A, Siller-Matula JM, Castriota F, Kubica J. Ticagrelor, but not clopidogrel and prasugrel, prevents ADP-induced vascular smooth muscle cell contraction: a placebo-controlled study in rats. Thromb Res. 2012 Jul;130(1):65-9. doi: 10.1016/j.thromres.2011.12.029. Epub 2012 Jan 21. PMID 22265722
- [Background] Saraste A, Nekolla S, Schwaiger M. Contrast-enhanced magnetic resonance imaging in the assessment of myocardial infarction and viability. J Nucl Cardiol. 2008 Jan-Feb;15(1):105-17. doi: 10.1007/BF02976902. Epub 2007 Dec 21. PMID 18242487
- [Background] Roes SD, Kelle S, Kaandorp TA, Kokocinski T, Poldermans D, Lamb HJ, Boersma E, van der Wall EE, Fleck E, de Roos A, Nagel E, Bax JJ. Comparison of myocardial infarct size assessed with contrast-enhanced magnetic resonance imaging and left ventricular function and volumes to predict mortality in patients with healed myocardial infarction. Am J Cardiol. 2007 Sep 15;100(6):930-6. doi: 10.1016/j.amjcard.2007.04.029. Epub 2007 Jul 5. PMID 17826372
- [Background] Bello D, Fieno DS, Kim RJ, Pereles FS, Passman R, Song G, Kadish AH, Goldberger JJ. Infarct morphology identifies patients with substrate for sustained ventricular tachycardia. J Am Coll Cardiol. 2005 Apr 5;45(7):1104-8. doi: 10.1016/j.jacc.2004.12.057. PMID 15808771
- [Background] Gudmundsson P, Winter R, Dencker M, Kitlinski M, Thorsson O, Ljunggren L, Willenheimer R. Real-time perfusion adenosine stress echocardiography versus myocardial perfusion adenosine scintigraphy for the detection of myocardial ischaemia in patients with stable coronary artery disease. Clin Physiol Funct Imaging. 2006 Jan;26(1):32-8. doi: 10.1111/j.1475-097X.2005.00646.x. PMID 16398668
- [Background] Stork A, Muellerleile K, Bansmann PM, Graessner J, Kaul M, Kemper J, Adam G, Lund GK. Value of T2-weighted, first-pass and delayed enhancement, and cine CMR to differentiate between acute and chronic myocardial infarction. Eur Radiol. 2007 Mar;17(3):610-7. doi: 10.1007/s00330-006-0460-6. Epub 2006 Dec 6. PMID 17149626
- [Background] Knopp MV, Schoenberg SO, Rehm C, Floemer F, von Tengg-Kobligk H, Bock M, Hentrich HR. Assessment of gadobenate dimeglumine for magnetic resonance angiography: phase I studies. Invest Radiol. 2002 Dec;37(12):706-15. doi: 10.1097/00004424-200212000-00011. PMID 12447005
- [Background] McCrohon JA, Moon JC, Prasad SK, McKenna WJ, Lorenz CH, Coats AJ, Pennell DJ. Differentiation of heart failure related to dilated cardiomyopathy and coronary artery disease using gadolinium-enhanced cardiovascular magnetic resonance. Circulation. 2003 Jul 8;108(1):54-9. doi: 10.1161/01.CIR.0000078641.19365.4C. Epub 2003 Jun 23. PMID 12821550
- [Background] Vohringer M, Mahrholdt H, Yilmaz A, Sechtem U. Significance of late gadolinium enhancement in cardiovascular magnetic resonance imaging (CMR). Herz. 2007 Mar;32(2):129-37. doi: 10.1007/s00059-007-2972-5. PMID 17401755
- [Background] Mahrholdt H, Wagner A, Judd RM, Sechtem U, Kim RJ. Delayed enhancement cardiovascular magnetic resonance assessment of non-ischaemic cardiomyopathies. Eur Heart J. 2005 Aug;26(15):1461-74. doi: 10.1093/eurheartj/ehi258. Epub 2005 Apr 14. PMID 15831557
- [Background] Weinsaft JW, Klem I, Judd RM. MRI for the assessment of myocardial viability. Cardiol Clin. 2007 Feb;25(1):35-56, v. doi: 10.1016/j.ccl.2007.02.001. PMID 17478239
- [Background] Sparrow P, Messroghli DR, Reid S, Ridgway JP, Bainbridge G, Sivananthan MU. Myocardial T1 mapping for detection of left ventricular myocardial fibrosis in chronic aortic regurgitation: pilot study. AJR Am J Roentgenol. 2006 Dec;187(6):W630-5. doi: 10.2214/AJR.05.1264. PMID 17114517
- [Background] Camici GG, Sudano I, Noll G, Tanner FC, Luscher TF. Molecular pathways of aging and hypertension. Curr Opin Nephrol Hypertens. 2009 Mar;18(2):134-7. doi: 10.1097/MNH.0b013e328326093f. PMID 19434051
- [Background] Werner N, Nickenig G. Endothelial progenitor cells in health and atherosclerotic disease. Ann Med. 2007;39(2):82-90. doi: 10.1080/07853890601073429. PMID 17453672
- [Background] Boulanger CM, Amabile N, Tedgui A. Circulating microparticles: a potential prognostic marker for atherosclerotic vascular disease. Hypertension. 2006 Aug;48(2):180-6. doi: 10.1161/01.HYP.0000231507.00962.b5. Epub 2006 Jun 26. No abstract available. PMID 16801490
- [Background] Quyyumi AA, Waller EK, Murrow J, Esteves F, Galt J, Oshinski J, Lerakis S, Sher S, Vaughan D, Perin E, Willerson J, Kereiakes D, Gersh BJ, Gregory D, Werner A, Moss T, Chan WS, Preti R, Pecora AL. CD34(+) cell infusion after ST elevation myocardial infarction is associated with improved perfusion and is dose dependent. Am Heart J. 2011 Jan;161(1):98-105. doi: 10.1016/j.ahj.2010.09.025. PMID 21167340
- [Background] Geisler T, Fekecs L, Wurster T, Chiribiri A, Schuster A, Nagel E, Miller S, Gawaz M, Stellos K, Bigalke B. Association of platelet-SDF-1 with hemodynamic function and infarct size using cardiac MR in patients with AMI. Eur J Radiol. 2012 Apr;81(4):e486-90. doi: 10.1016/j.ejrad.2011.06.019. Epub 2011 Jul 2. PMID 21724347
- [Background] Sibbing D, Braun S, Morath T, Mehilli J, Vogt W, Schomig A, Kastrati A, von Beckerath N. Platelet reactivity after clopidogrel treatment assessed with point-of-care analysis and early drug-eluting stent thrombosis. J Am Coll Cardiol. 2009 Mar 10;53(10):849-56. doi: 10.1016/j.jacc.2008.11.030. PMID 19264241
- [Background] Gori T, Muxel S, Damaske A, Radmacher MC, Fasola F, Schaefer S, Schulz A, Jabs A, Parker JD, Munzel T. Endothelial function assessment: flow-mediated dilation and constriction provide different and complementary information on the presence of coronary artery disease. Eur Heart J. 2012 Feb;33(3):363-71. doi: 10.1093/eurheartj/ehr361. Epub 2011 Sep 14. PMID 21920964
- [Background] Spiro JR, Digby JE, Ghimire G, Mason M, Mitchell AG, Ilsley C, Donald A, Dalby MC, Kharbanda RK. Brachial artery low-flow-mediated constriction is increased early after coronary intervention and reduces during recovery after acute coronary syndrome: characterization of a recently described index of vascular function. Eur Heart J. 2011 Apr;32(7):856-66. doi: 10.1093/eurheartj/ehq401. Epub 2010 Oct 29. PMID 21037253
- [Background] Eshtehardi P, Windecker S, Cook S, Billinger M, Togni M, Garachemani A, Meier B, Hess OM, Wenaweser P. Dual low response to acetylsalicylic acid and clopidogrel is associated with myonecrosis and stent thrombosis after coronary stent implantation. Am Heart J. 2010 May;159(5):891-898.e1. doi: 10.1016/j.ahj.2010.02.025. PMID 20435201
- [Background] Breet NJ, van Werkum JW, Bouman HJ, Kelder JC, Ruven HJ, Bal ET, Deneer VH, Harmsze AM, van der Heyden JA, Rensing BJ, Suttorp MJ, Hackeng CM, ten Berg JM. Comparison of platelet function tests in predicting clinical outcome in patients undergoing coronary stent implantation. JAMA. 2010 Feb 24;303(8):754-62. doi: 10.1001/jama.2010.181. PMID 20179285
- [Background] Libby P, Ridker PM, Hansson GK; Leducq Transatlantic Network on Atherothrombosis. Inflammation in atherosclerosis: from pathophysiology to practice. J Am Coll Cardiol. 2009 Dec 1;54(23):2129-38. doi: 10.1016/j.jacc.2009.09.009. PMID 19942084
- [Background] Hansson GK, Hermansson A. The immune system in atherosclerosis. Nat Immunol. 2011 Mar;12(3):204-12. doi: 10.1038/ni.2001. PMID 21321594
- [Background] Libby P, Ridker PM, Hansson GK. Progress and challenges in translating the biology of atherosclerosis. Nature. 2011 May 19;473(7347):317-25. doi: 10.1038/nature10146. PMID 21593864
- [Background] Hofmann U, Beyersdorf N, Weirather J, Podolskaya A, Bauersachs J, Ertl G, Kerkau T, Frantz S. Activation of CD4+ T lymphocytes improves wound healing and survival after experimental myocardial infarction in mice. Circulation. 2012 Apr 3;125(13):1652-63. doi: 10.1161/CIRCULATIONAHA.111.044164. Epub 2012 Mar 2. PMID 22388323
- [Background] Bernal-Mizrachi L, Jy W, Jimenez JJ, Pastor J, Mauro LM, Horstman LL, de Marchena E, Ahn YS. High levels of circulating endothelial microparticles in patients with acute coronary syndromes. Am Heart J. 2003 Jun;145(6):962-70. doi: 10.1016/S0002-8703(03)00103-0. PMID 12796750
- [Background] Kyaw T, Tipping P, Toh BH, Bobik A. Current understanding of the role of B cell subsets and intimal and adventitial B cells in atherosclerosis. Curr Opin Lipidol. 2011 Oct;22(5):373-9. doi: 10.1097/MOL.0b013e32834adaf3. PMID 21881498
- [Background] Kyaw T, Tay C, Hosseini H, Kanellakis P, Gadowski T, MacKay F, Tipping P, Bobik A, Toh BH. Depletion of B2 but not B1a B cells in BAFF receptor-deficient ApoE mice attenuates atherosclerosis by potently ameliorating arterial inflammation. PLoS One. 2012;7(1):e29371. doi: 10.1371/journal.pone.0029371. Epub 2012 Jan 4. PMID 22238605
- [Background] Martin JC, Canlet C, Delplanque B, Agnani G, Lairon D, Gottardi G, Bencharif K, Gripois D, Thaminy A, Paris A. 1H NMR metabonomics can differentiate the early atherogenic effect of dairy products in hyperlipidemic hamsters. Atherosclerosis. 2009 Sep;206(1):127-33. doi: 10.1016/j.atherosclerosis.2009.01.040. Epub 2009 Feb 7. PMID 19324361
- [Background] Lewis GD, Asnani A, Gerszten RE. Application of metabolomics to cardiovascular biomarker and pathway discovery. J Am Coll Cardiol. 2008 Jul 8;52(2):117-23. doi: 10.1016/j.jacc.2008.03.043. PMID 18598890
- [Background] Watson AD. Thematic review series: systems biology approaches to metabolic and cardiovascular disorders. Lipidomics: a global approach to lipid analysis in biological systems. J Lipid Res. 2006 Oct;47(10):2101-11. doi: 10.1194/jlr.R600022-JLR200. Epub 2006 Aug 10. PMID 16902246
- [Background] Lewis GD, Wei R, Liu E, Yang E, Shi X, Martinovic M, Farrell L, Asnani A, Cyrille M, Ramanathan A, Shaham O, Berriz G, Lowry PA, Palacios IF, Tasan M, Roth FP, Min J, Baumgartner C, Keshishian H, Addona T, Mootha VK, Rosenzweig A, Carr SA, Fifer MA, Sabatine MS, Gerszten RE. Metabolite profiling of blood from individuals undergoing planned myocardial infarction reveals early markers of myocardial injury. J Clin Invest. 2008 Oct;118(10):3503-12. doi: 10.1172/JCI35111. PMID 18769631
- [Background] Zhang F, Jia Z, Gao P, Kong H, Li X, Chen J, Yang Q, Yin P, Wang J, Lu X, Li F, Wu Y, Xu G. Metabonomics study of atherosclerosis rats by ultra fast liquid chromatography coupled with ion trap-time of flight mass spectrometry. Talanta. 2009 Aug 15;79(3):836-44. doi: 10.1016/j.talanta.2009.05.010. Epub 2009 May 19. PMID 19576453
- [Background] Mayr M, Chung YL, Mayr U, Yin X, Ly L, Troy H, Fredericks S, Hu Y, Griffiths JR, Xu Q. Proteomic and metabolomic analyses of atherosclerotic vessels from apolipoprotein E-deficient mice reveal alterations in inflammation, oxidative stress, and energy metabolism. Arterioscler Thromb Vasc Biol. 2005 Oct;25(10):2135-42. doi: 10.1161/01.ATV.0000183928.25844.f6. Epub 2005 Aug 25. PMID 16123314
- [Background] Li N, Liu JY, Timofeyev V, Qiu H, Hwang SH, Tuteja D, Lu L, Yang J, Mochida H, Low R, Hammock BD, Chiamvimonvat N. Beneficial effects of soluble epoxide hydrolase inhibitors in myocardial infarction model: Insight gained using metabolomic approaches. J Mol Cell Cardiol. 2009 Dec;47(6):835-45. doi: 10.1016/j.yjmcc.2009.08.017. Epub 2009 Aug 28. PMID 19716829
- [Background] Liu JY, Yang J, Inceoglu B, Qiu H, Ulu A, Hwang SH, Chiamvimonvat N, Hammock BD. Inhibition of soluble epoxide hydrolase enhances the anti-inflammatory effects of aspirin and 5-lipoxygenase activation protein inhibitor in a murine model. Biochem Pharmacol. 2010 Mar 15;79(6):880-7. doi: 10.1016/j.bcp.2009.10.025. Epub 2009 Nov 5. PMID 19896470
- [Background] Ferreira CR, Saraiva SA, Catharino RR, Garcia JS, Gozzo FC, Sanvido GB, Santos LF, Lo Turco EG, Pontes JH, Basso AC, Bertolla RP, Sartori R, Guardieiro MM, Perecin F, Meirelles FV, Sangalli JR, Eberlin MN. Single embryo and oocyte lipid fingerprinting by mass spectrometry. J Lipid Res. 2010 May;51(5):1218-27. doi: 10.1194/jlr.D001768. Epub 2009 Nov 5. PMID 19965589
- [Background] Saric J, Want EJ, Duthaler U, Lewis M, Keiser J, Shockcor JP, Ross GA, Nicholson JK, Holmes E, Tavares MF. Systematic evaluation of extraction methods for multiplatform-based metabotyping: application to the Fasciola hepatica metabolome. Anal Chem. 2012 Aug 21;84(16):6963-72. doi: 10.1021/ac300586m. Epub 2012 Aug 10. PMID 22799605
- [Background] Caricilli AM, Picardi PK, de Abreu LL, Ueno M, Prada PO, Ropelle ER, Hirabara SM, Castoldi A, Vieira P, Camara NO, Curi R, Carvalheira JB, Saad MJ. Gut microbiota is a key modulator of insulin resistance in TLR 2 knockout mice. PLoS Biol. 2011 Dec;9(12):e1001212. doi: 10.1371/journal.pbio.1001212. Epub 2011 Dec 6. PMID 22162948 (Retraction: PMID 27213533 Caricilli AM, Picardi PK, de Abreu LL, Ueno M, Prada PO, Ropelle ER, Hirabara SM, Castoldi Â, Vieira P, Camara NO, Curi R, Carvalheira JB, Saad MJ. PLoS Biol. 2016 May;14(5):e1002479)
- [Background] Wang J, Ruotsalainen S, Moilanen L, Lepisto P, Laakso M, Kuusisto J. The metabolic syndrome predicts cardiovascular mortality: a 13-year follow-up study in elderly non-diabetic Finns. Eur Heart J. 2007 Apr;28(7):857-64. doi: 10.1093/eurheartj/ehl524. Epub 2007 Feb 15. PMID 17303589
- [Background] Vamos EP, Millett C, Parsons C, Aylin P, Majeed A, Bottle A. Nationwide study on trends in hospital admissions for major cardiovascular events and procedures among people with and without diabetes in England, 2004-2009. Diabetes Care. 2012 Feb;35(2):265-72. doi: 10.2337/dc11-1682. Epub 2011 Dec 30. PMID 22210568
- [Background] Nicolau JC, Serrano CV Jr, Giraldez RR, Baracioli LM, Moreira HG, Lima F, Franken M, Kalil R, Ramires JA, Giugliano RP. In patients with acute myocardial infarction, the impact of hyperglycemia as a risk factor for mortality is not homogeneous across age-groups. Diabetes Care. 2012 Jan;35(1):150-2. doi: 10.2337/dc11-1170. Epub 2011 Oct 25. PMID 22028280
- [Background] Hattori M, Taylor TD. The human intestinal microbiome: a new frontier of human biology. DNA Res. 2009 Feb;16(1):1-12. doi: 10.1093/dnares/dsn033. Epub 2009 Jan 15. PMID 19147530
- [Background] de Kort S, Keszthelyi D, Masclee AA. Leaky gut and diabetes mellitus: what is the link? Obes Rev. 2011 Jun;12(6):449-58. doi: 10.1111/j.1467-789X.2010.00845.x. Epub 2011 Mar 8. PMID 21382153
- [Derived] Fonseca FA, Caixeta A, Szarf G, Pinto I, Figueiredo Neto AM, Franca CN, Bianco HT, Fonseca HA, Bacchin AS, Birtche M, Batista IRM, Izar MC; BATTLE-AMI investigators. Smaller infarct size with ticagrelor vs. clopidogrel in STEMI patients: Insights from cardiac magnetic resonance. PLoS One. 2025 Oct 27;20(10):e0328114. doi: 10.1371/journal.pone.0328114. eCollection 2025. PMID 41144431
- [Derived] da Silva LS, Germano DB, Fonseca FAH, Shio MT, da Silva Nali LH, Tuleta ID, Juliano Y, de Oliveira Izar MC, Ribeiro AP, Kato JT, do Amaral JB, Franca CN. Persistence of a proinflammatory status after treatment of the acute myocardial infarction. Geriatr Gerontol Int. 2023 Sep;23(9):700-707. doi: 10.1111/ggi.14649. Epub 2023 Jul 31. PMID 37522226
- [Derived] Lotfollahi Z, Mello APQ, Fonseca FAH, Machado LO, Mathias AF, Izar MC, Damasceno NRT, Oliveira CLP, Neto AMF. Changes in lipoproteins associated with lipid-lowering and antiplatelet strategies in patients with acute myocardial infarction. PLoS One. 2022 Aug 30;17(8):e0273292. doi: 10.1371/journal.pone.0273292. eCollection 2022. PMID 36040917
- [Derived] Pinto LCS, Mello APQ, Izar MCO, Damasceno NRT, Neto AMF, Franca CN, Caixeta A, Bianco HT, Povoa RMS, Moreira FT, Bacchin ASF, Fonseca FA. Main differences between two highly effective lipid-lowering therapies in subclasses of lipoproteins in patients with acute myocardial infarction. Lipids Health Dis. 2021 Sep 29;20(1):124. doi: 10.1186/s12944-021-01559-w. PMID 34587943
- [Derived] Klassen A, Faccio AT, Picossi CRC, Derogis PBMC, Dos Santos Ferreira CE, Lopes AS, Sussulini A, Cruz ECS, Bastos RT, Fontoura SC, Neto AMF, Tavares MFM, Izar MC, Fonseca FAH. Evaluation of two highly effective lipid-lowering therapies in subjects with acute myocardial infarction. Sci Rep. 2021 Aug 5;11(1):15973. doi: 10.1038/s41598-021-95455-z. PMID 34354179
- [Derived] Fonseca FAH, Izar MC, Maugeri IML, Berwanger O, Damiani LP, Pinto IM, Szarf G, Franca CN, Bianco HT, Moreira FT, Caixeta A, Alves CMR, Soriano Lopes A, Klassen A, Tavares MFM, Fonseca HA, Carvalho ACC; BATTLE-AMI Investigators. Effects of four antiplatelet/statin combined strategies on immune and inflammatory responses in patients with acute myocardial infarction undergoing pharmacoinvasive strategy: Design and rationale of the B and T Types of Lymphocytes Evaluation in Acute Myocardial Infarction (BATTLE-AMI) study: study protocol for a randomized controlled trial. Trials. 2017 Dec 19;18(1):601. doi: 10.1186/s13063-017-2361-1. PMID 29258572